CLINICAL TRIAL: NCT07305805
Title: A Multiple Dose Study Investigating Pharmacodynamics and Pharmacokinetics of Subcutaneous NNC0363-1063 in Participants With Type 1 Diabetes
Brief Title: A Research Study of a New Medicine NNC0363-1063 in Participants With Type 1 Diabetes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1644-8194; U1111-1317-2815 (Other: World Health Organization (WHO)); 2025-521593-33 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): Participants will receive NNC0363-1063 co-administered with and without non-glucose carbohydrate in treatment period 1 and treatment period 2.
  Interventions: Drug: NNC0363-1063
- Sequence 2 (Experimental): Participants will receive NNC0363-1063 co-administered with and without non-glucose carbohydrate in treatment period 1 and treatment period 2.
  Interventions: Drug: NNC0363-1063
- Sequence 3 (Experimental): Participants will receive NNC0363-1063 co-administered with and without non-glucose carbohydrate in treatment period 1 and treatment period 2.
  Interventions: Drug: NNC0363-1063
- Sequence 4 (Experimental): Participants will receive NNC0363-1063 co-administered with and without non-glucose carbohydrate in treatment period 1 and treatment period 2.
  Interventions: Drug: NNC0363-1063

INTERVENTIONS:
Drug: NNC0363-1063 — NNC0363-1063 will be administered subcutaneously.

SUMMARY:
The purpose of this clinical study is to find out how the novel insulin NNC0363-1063 and a non-glucose carbohydrate used in food and beverage might interact in participants with type 1 diabetes and if co-administration of these substances is safe and tolerable. All participants will get a fixed dose of NNC0363-1063 and an oral administration of different amounts of the non-glucose carbohydrate in a random order during 4 interaction tests. The participants will be in this clinical study for about 5 to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant (sex at birth) of non-child bearing potential. Non-child bearing potential being defined as surgically sterilised (i.e., documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or being postmenopausal (defined as no menses for 12 month without an alternative medical cause) prior to the day of screening.
* Age 18-64 years (both inclusive) at the time of signing informed consent.
* Body mass index between 18.5-29.9 Kilogram Per Square Meter (kg/m^2) (both inclusive) at the day of screening.
* Diagnosed with type 1 diabetes mellitus greater than or equal to (≥) 1 year prior to the day of screening.
* Treated with multiple daily insulin injections or continuous subcutaneous insulin infusion ≥ 90 days prior to the day of screening.
* Glycated haemoglobin (HbA1c) less than or equal to (≤ ) 9.0 percentage (%) at the day of screening.

Exclusion Criteria:

* Male of reproductive age who, or whose female partner(s), is not using an adequate contraceptive method.
* Any condition, except for mild conditions under stable treatment associated with type 1 diabetes mellitus, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-05-17 (Estimated); Study Completion 2026-05-21 (Estimated)

PRIMARY OUTCOMES:
AUC, GIR,SS: Area under the glucose infusion rate-time curve at steady state | Visit 2 and 3: Day 2 and 3
  Measured in milligrams per kilogram (mg/kg).

SECONDARY OUTCOMES:
GIRmax,SS: Maximum glucose infusion rate at steady state | Visit 2 and 3: Day 2 and 3
  Measured in milligrams per kilogram*minute (mg/[kg*min]).
Time to maximum glucose infusion rate (tGIRmax),SS: Time to maximum glucose infusion rate at steady state | Visit 2 and 3: Day 2 and 3
  Measured in hours.
AUC,I1063,SS: Area under the serum NNC0363-1063 concentration time curve at steady state | Visit 2 and 3: Day 2 and 3
  Measured in hours*picomoles per litre (h*pmol/L).
Cmax,I1063,SS: Maximum observed serum NNC0363-1063 concentration at steady state | Visit 2 and 3: Day 2 and 3
  Measured in picomoles per litre (pmol/L).
tmax,I1063,SS: Time to maximum observed serum NNC0363-1063 concentration at steady state | Visit 2 and 3: Day 2 and 3
  Measured in hours.
Number of adverse events | Visit 2 and 3: Day 2 and 3
  Measured as number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com